CLINICAL TRIAL: NCT07401667
Title: Efficacy of Connective Tissue Graft Versus Titanium Papillary Inserts in the Surgical Reconstruction of Interdental Papilla
Brief Title: Comparison of Connective Tissue Graft Versus Titanium Papillary Inserts in the Surgical Reconstruction of Interdental Papilla.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr R Viswa Chandra (Other)
Collaborators: SVS Institute of Dental Sciences (Other)
Responsible Party: Sponsor-Investigator, Dr R Viswa Chandra, PROFESSOR AND HEAD OF DEPARTMENT, SVS Institute of Dental Sciences
Organization: SVS Institute of Dental Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SVSIDS/PERIO/4/2022
Record Dates: First submitted 2025-08-30; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Papilla Reconstruction
Keywords: Connective tissue grafts; titanium inserts; black triangle; papilla height; papilla reconstruction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TITANIUM INSERTS FOR PAPILLA RECONSTRUCTION (Experimental)
  Interventions: Device: TITANIUM INSERTS
- SUB-EPITHELIAL CONNECTIVE TISSUE GRAFT FOR PAPILLA RECONSTRUCTION USING HAN & TAKEI TECHNIQUE (Active Comparator)
  Interventions: Procedure: CONNECTIVE TISSUE GRAFT

INTERVENTIONS:
Device: TITANIUM INSERTS — The titanium papillary insert2 is composed of a pyramidal- shaped polished titanium core; it has a height of 2 to 3 mm and a base that is 3 mm bucco-lingually and 1 mm in the mesio-distal dimension. It also has mesial and distal concavities to allow for the emergence of the papilla. It is fitted into the bone between two adjacent teeth by means of a self-taping screw extension that is 0.8 mm in diameter and 5 mm in length.
  Arms: TITANIUM INSERTS FOR PAPILLA RECONSTRUCTION
Procedure: CONNECTIVE TISSUE GRAFT — CTG is widely used across a broad range of clinical indications in periodontal and peri-implant therapy. It is primarily indicated for the treatment of gingival recession, reduction of dentinal hypersensitivity, and correction of mucogingival deformities.
  Arms: SUB-EPITHELIAL CONNECTIVE TISSUE GRAFT FOR PAPILLA RECONSTRUCTION USING HAN & TAKEI TECHNIQUE

SUMMARY:
Aim and Objectives: The study aimed to evaluate the effectiveness of titanium inserts for interdental papilla reconstruction, comparing it with the Han and Takei technique using subepithelial connective tissue grafts. The objectives included assessing the black triangle height, papilla height and papilla presence index (PPI) at baseline, 1 month and 3 months post operatively along with the evaluation of Early Wound Healing Score (EHS) during the first week of post operative healing period. Patients and Methods: This single-blind randomized clinical trial included systemically healthy individuals aged 18-35 years with Nordland and Tarnow's Class I-III papillary loss. A total of 18 participants were randomly assigned to either test group or control group. Clinical parameters were measured pre- and post-operatively at specified intervals. Both groups received standard presurgical care and postoperative follow-up. The surgical protocol for the test group involved titanium insert placement in the interdental bone, while the control group received a connective tissue graft using the Han and Takei method.

DETAILED DESCRIPTION:
INTRODUCTION The human gingiva consists of specific anatomical components: the attached gingiva, which securely connects the gingiva to the underlying bone, and the marginal (free) gingiva, a slender strip of tissue that surrounds the tooth without adhering to hard tissue. Vertically, the marginal gingiva stretches from the (Cemento-enamel junction) CEJ to the free gingival groove. In the interdental space lies the interdental papilla, a vital part of the gingival structure.1,2 Morphologically, the interdental papilla reaches from the interdental alveolar bone to the contact point of neighboring teeth. It is separated from the mesial and distal aspects by sulcular and/or junctional epithelium, whereas the facial and oral surfaces are covered by keratinized gingival oral epithelium. The development of the interdental papilla takes place during tooth eruption, and its shape is affected by the contact points of neighboring teeth, the widths of proximal tooth surfaces, and the configuration of the CEJ.1,2 The interdental papilla can be vulnerable to inflammatory agents through the junctional/sulcular epithelia, leading to localized inflammation even in clinically healthy papillae, which is a frequently observed histologic finding.

A black triangle, which denotes the loss of interdental papillae, continues to be one of the most prevalent conditions leading to not just aesthetic and phonetic issues but also functional challenges as it increases the likelihood of food impaction that negatively impacts periodontal health. The interdental papilla in the incisor area is typically pyramidal in form. Elements that affect the presence or absence of interdental papilla include crestal alveolar bone height, the dimensions of the interproximal space, soft tissue appearance (thick or thin biotype), buccal plate thickness, the type of contact area (triangular versus square), and the biologic width.3 The limited ability of the interdental papilla to regenerate seems to be influenced by various aspects, such as anatomical factors, bone loss, plaque accumulation, and inflammatory phenomena within the interdental area. Moreover, there is an indication that the interdental papilla may have unique functional features resulting from specific cellular or molecular attributes. This idea is supported by ample documentation showing that distinct anatomical tissue units, even within the marginal gingiva, display specific characteristics. 4-9 A range of techniques has been investigated for reconstructing the interdental papilla, encompassing both nonsurgical and surgical strategies. Among the nonsurgical techniques are repeated curettage of the interdental papilla, orthodontic adjustments, restorative fixes, and the application of hyaluronic acid (HA). Although these methods have been tried, they frequently produce less reliable results and provide limited potential for considerable papilla enhancement.

Conversely, surgical approaches have become more prominent due to their effectiveness in papilla reconstruction, despite being more invasive and complex. These surgical options consist of pedicle and free gingival grafts, connective tissue grafts (CTG), subepithelial connective tissue grafts (SCTG), and the application of Choukroun's platelet-rich fibrin (PRF). These techniques involve the manipulation of gum tissues to improve the height and shape of the interdental papilla, targeting more reliable and satisfactory aesthetic results.10 Titanium alloys are highly regarded for their outstanding strength-to-weight ratio, resistance to corrosion, and biocompatibility, which makes them suitable for aerospace, medical implants, and marine uses. Their ability to resist oxygen, water, and chemicals guarantees durability in harsh conditions, while their non-toxic nature makes them ideal for medical applications. The characteristics of titanium alloys can be customized through alloying, heat treatment, and surface modifications to satisfy specific application demands.11 El Askary et al (2000)12 described the papillary titanium insert and emphasized its benefits, manipulation, and handling. To support the soft tissue between two implants and achieve the desired interdental papilla-like form, a papillary titanium insert was created. This method eliminates the necessity for any bone grafting procedures while requiring fewer tools and reducing the number of surgical interventions.

This study seeks to present the use of a titanium insert for reconstructing the interdental papilla, which was previously utilized by El Askary et al12 for forming inter-implant papillae. It also intends to compare this method with the Han and Takei technique13 of papilla reconstruction using a subepithelial connective tissue graft. The research findings hold the potential to provide clinicians with an innovative therapeutic alternative for enhancing periodontal aesthetics and increasing patient satisfaction.

MATERIAL AND METHODS

TRIAL DESIGN:

The trial was designed as a single-blind randomized controlled clinical trial to clinically evaluate the use of a titanium insert and subepithelial connective tissue graft for the reconstruction of Interdental papilla.

PARTICIPANTS AND ELIGIBILITY CRITERIA:

Subjects for the study were selected from the outpatient section of the Department of Periodontology, Sri Venkata Sai Institute of Dental Sciences, Mahabubnagar, Telangana and were followed up over three months period after the procedures. The design of the research was approved by Institutional Ethics Committee with approval number SVSIDS/Perio/2/2022. Systemically healthy male and female patients with a stable periodontal health of age 18-35 years. Patients with Nordland and Tarnow's13 Class I, II, III interdental papillary loss at a single site and Gingival recession <2 mm on the facial aspect. Patients presenting with adequate width of attached gingiva (2-3mm) and having a thick gingival biotype (2 mm) were included into the study. Midline diastema patients, medically compromised patients, Pregnant and lactating women, heavy smokers, patient who underwent radiotherapy & chemotherapy, patients with any bleeding or clotting disorders and patients not willing to participate in the study were not included into the study.

SAMPLE SIZE CALCULATION:

Assuming an anticipated prevalence of 36.42%, the necessary sample size is 18 to achieve a margin of error or absolute accuracy of +25% in the prevalence prediction with 95% confidence, taking into account a possible loss or attrition of 15%. At this sample size, the expected 95% CI is 11. 42%. The Scalex SP calculator (Naing L, et. al., 2022) is used to determine this sample size.

RANDOMIZATION AND BLINDING:

In order to assess the effectiveness of "Titanium inserts" in interdental papilla augmentation procedures, the experiment was set up as a randomized controlled clinical trial with single blinding. Randomization included the use of a computer to generate the allocation sequence in random permuted blocks (block randomization), and blinding was achieved by having a second operator assign the block of sites to study groups according to the sequence by which the first operator had coded the two treatment sites selected from each patient into the following groups. Titanium inserts for interdental papilla reconstruction (test group) and connective tissue graft for interdental papilla reconstruction (control group). Until this clinical experiment was over, the blind was not breached.

INTERVENTIONS:

Pre-Surgical Protocol:

The first phase of treatment for each patient included scaling and root planning, occlusal adjustment, and oral hygiene education in preparation for the procedure. Following the initial examination and thorough phase I treatment, the patients were reevaluated one week later to determine whether they had maintained their oral hygiene. After two weeks, the patients were brought back for the operation.

Study Protocol:

Before the operation, all baseline parameters (measured on the day of the surgery) were recorded. The following variables were noted: interdental papilla height, Black triangle height, and PPI, which was calculated by Cardaropoli et al.15, at baseline and again one month and three months after the procedure. The EHS developed by Marini et al.16 was used one week after surgery to evaluate soft tissue wound healing. All measurements are taken to the closest millimeter.

SURGICAL PROCEDURE:

In Test Site:

After rinsing with an antiseptic solution for one-minute, adequate amount of local anesthesia was administered. Using a 15C blade, a crevicular incision was made around each tooth, with no incisions across the interdental papilla. Horizontal incision was made at the base of the papilla on the buccal side of the adjacent teeth. Two vertical relaxing incisions were made, parallel to line angle of the adjacent tooth on either side. Semilunar incision was made at the base of the papilla on the palatal side of the interdental space that is to be reconstructed. A full thickness flap was raised apically and the preserved papilla is then elevated with an Orban knife or curettes, intact to the remaining facial flap. After reflection of flap, at the recipient site, a 1-mm diameter twist drill is used to drill midway between the two teeth to a depth of 5 mm. The insert is grasped with pliers and threaded into the osteotomy until it is completely flush with the bone crest which allows for the protrusion of the papilla core of the insert. Soft tissue closure is then achieved through relaxing incisions, and the stripping of the periosteum at the base of the flap allows for a tension- free closure.

In Control Site:

After rinsing with an antiseptic solution for one-minute, adequate amount of local anesthesia was administered. Han and Takei technique13 using subepithelial connective tissue graft was planned to be performed. Using a 15-no. blade was used to make a semilunar incision from the disto-labial line angle to the mesio-labial line angle of tooth, at a distance of 6-10 mm in the apical direction from the marginal gingiva in the interdental region. A 12-no. blade was used to make intrasulcular incisions around the mesial half and the distal half of the two adjacent teeth. The gingival-papillary unit was pushed incisally to move gingiva into the crated area to create a split-thickness pouch. The interdental papillary unit was coronally advanced. Subepithelial connective tissue double the size of missing papillary height was harvested from palate. The connective tissue was placed into the pouch space. The semilunar incision was sutured with the interrupted suture, whereas the gingival-papillary unit was sutured coronally using suspensory suture technique.

POSTSURGICAL CARE:

For both the groups, routine postsurgical instructions were given and systemic antibiotics (Amoxicillin-Clavulanate Potassium 625mg thrice daily) was prescribed for 3 days and analgesic (Ibuprofen 800 mg twice daily) for 3 days. A rinse with 10 ml of 0.12% chlorhexidine mouthwash twice daily for 2 weeks was recommended for all the patients. Patients were advised to refrain using any interdental cleansing aids for 4 weeks. Patients were recalled at the end of 1 week for the removal of sutures and every month for oral hygiene maintenance. Clinical measurements were repeated after 1 month and 3-month interval.

OUTCOMES:

Primary outcomes:

Interdental papilla height:

It is to be measured from base of the papilla (a line joining the two adjacent teeth gingival zenith) to the tip of the papilla using a UNC-15 probe.

Black triangle height:

It is to be measured from the tip of the interdental papilla to the apical-most point of the contact point using a UNC-15 probe Papilla presence index (PPI) given by Cardaropoli et al: 15 The classification system presented here is based on the positional relationship among the papilla, CEJ, and adjacent teeth.

Papilla Presence Index score 1 (PPI 1) is reported when the papilla is completely present and coronally extends to the contact point to completely fill the inter- proximal embrasure. This papilla is at the same level as the adjacent papillae.

Papilla Presence Index score 2 (PPI 2) describes a papilla that is no longer completely present and lies apical to the contact point. This papilla is not at the same level as the adjacent papillae, and the embrasure is no longer completely filled, but the iCEJ is still not visible.

Both PPI 1 and PPI 2 scores can be complicated by the presence of buccal gingival recession, classified as PPI 1r and PPI 2r.

Papilla Presence Index score 3 (PPI 3) refers to the situation in which the papilla is moved more apical and the iCEJ becomes visible. This situation is compatible with a great amount of interdental soft tissue recession.

Papilla Presence Index score 4 (PPI 4) describes when the papilla lies apical to both the iCEJ and buccal CEJ (bCEJ). Interproximal soft tissue recession is present together with buccal gingival recession, and patient esthetics is dramatically compromised.

Secondary Outcome:

Postoperatively after 1-week, soft tissue wound healing will be assessed by using Early Wound Healing Score (EHS) by Marini et al16. The EHS scoring was based on the evaluation of clinical signs of re-epithelialization, hemostasis and inflammation. The sum of the single scores for these three parameters calculates the EHS, which ranges between 0 to 10 points.

STATISTICAL ANALYSIS The data was analyzed using SPSS© version 22 (IBM, India). Friedman test is used to compare the parameters at various intervals, Post hoc analysis using Bonferroni calculations were used for intra group comparisons and Mann-Whitney U test was used for the inter group comparison of parameters. p value less than 0.05 was set as significant and a value lesser than 0.001 was highly significant.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy male and female patients with a stable periodontal health of age 18-35 years.
* Patients with Nordland and Tarnow's1 Class I, II, III interdental papillary loss at a single site and Gingival recession < 2 mm on the facial aspect.
* Patients presenting with adequate width of attached gingiva (2-3mm)
* Having a thick gingival biotype (2 mm)

Exclusion Criteria:

* Midline diastema patients
* Medically compromised patients
* Pregnant and lactating women
* Heavy smokers,
* Patient who underwent radiotherapy & chemotherapy,
* Patients with any bleeding or clotting disorders
* Patients not willing to participate in the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-05-21 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Interdental papilla height | 3 MONTHS
  To be measured from base of the papilla (a line joining the two adjacent teeth gingival zenith) to the tip of the papilla. Measured with UNC-15 probe.
Black triangle height | 3 MONTHS
  Measurement from the tip of the interdental papilla to the apical-most point of the contact point. Measured using a digital vernier caliper.
Papilla presence index (PPI) | 3 MONTHS
  given by Cardaropoli et al

SECONDARY OUTCOMES:
Early Wound Healing Score (EHS) | 1 WEEK
  GIVEN BY Lorenzo Marini

CONTACTS AND LOCATIONS:
Locations (1):
- Svs Institute of Dental Sciences, Mahbūbnagar, Telangana, India

IPD SHARING:
Plan to Share IPD: Yes